CLINICAL TRIAL: NCT07265739
Title: A Phase 2 Study of Losartan in Combination With Weekly Paclitaxel in Platinum Resistant Ovarian Cancer
Brief Title: Losartan and Paclitaxel in Platinum Resistant Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Oladapo O. Yeku,M.D.,Ph.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-680
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Platinum Resistant Ovarian Cancer
Keywords: Platinum Resistant Ovarian Cancer; epithelial ovarian carcinoma; fallopian tube carcinoma; primary peritoneal carcinoma
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Losartan; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Losartan + Paclitaxel (Experimental): Once daily oral losartan combined with paclitaxel administered intravenously once weekly. Each cycle is 21 days and participants may receive study treatment until disease progression or withdrawal. Losartan and paclitaxel are administered at a pre-determined dose.
  Interventions: Drug: losartan; Drug: Paclitaxel

INTERVENTIONS:
Drug: losartan — Treatment with losartan will be administered orally once daily starting on day 1 of every 21-day cycle and will be taken continuously throughout the cycle. Losartan is administered at 25 mg a day for the first 7 days of cycle 1. Losartan may be increased to 50 mg daily on day 8 if systolic blood pressure ≥ 120 mm Hg.
Drug: Paclitaxel — Paclitaxel 80 mg/m2 will be administered as a 60-min intravenous infusion after any premedication as per institutional guidelines. A ramp-up infusion rate is also acceptable as per institutional guidelines. Paclitaxel will be administered on days 1, 8 and 15 of a 21-day cycle and treatment will continue until unacceptable toxicity or disease progression.

SUMMARY:
The purpose of this Phase II study is to measure the effects of a combination of study drugs, losartan and paclitaxel, on platinum resistant ovarian cancer.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open label study of daily oral losartan in combination with intravenous weekly paclitaxel in patients with platinum resistant ovarian cancer. The primary endpoint of this study is overall response rate (ORR) and the secondary endpoint is progression free survival.

The U.S. Food and Drug Administration (FDA) has not approved losartan for this specific disease but it has been approved for other uses. The U.S. Food and Drug Administration (FDA) has approved paclitaxel as a treatment option for this disease. This research study involves screening for eligibility, study treatment with the study drugs, and study visits. Participants will receive study treatment until disease progression, withdrawal, or unacceptable side effects are experienced. Participants that stop study treatment due to disease progression will be followed for 30 days. Participants that stop study treatment due to an unacceptable side effect will have visits and imaging scans every 9 weeks until a different treatment is started. It is expected that about 27 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 18 years of age.
* Subjects with histologically/cytologically confirmed advanced epithelial ovarian, fallopian tube, or primary peritoneal carcinoma. Subjects with mucinous carcinoma and low-grade serous carcinoma are not eligible.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥20 mm (≥2 cm) by chest x-ray or as ≥10 mm (≥1 cm) with CT scan, MRI, or calipers by clinical exam.
* Subject is able to provide written, informed consent before initiation of any study related procedures, and is able, in the opinion of the investigator, to comply with all the requirements of the study.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Subject has adequate organ function at screening:

  i) absolute neutrophil count (ANC) ≥ 1000/mm3 without the use of hematopoietic growth factors.

ii) platelet count ≥ 75,000/mm3. iii) hemoglobin ≥ 8.0 g/dL (must be at least 1 weeks post-red blood cell transfusion and not receiving erythropoietic-stimulating agents).

iv) total bilirubin ≤ 1.5 × the upper limit of normal (ULN). For subjects with documented Gilbert's disease, total bilirubin ≤ 3.0 mg/dL is allowed.

v) serum albumin ≥ 2.5 g/dL vi) serum creatinine clearance (CrCl) ≥ 40 mL/min, using Cockcroft and Gault vii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN in the absence of documented liver metastases; ≤ 5 x ULN in the presence of liver metastases.

* Prior to study Day 1 (first study treatment administration), subject must be:

  i) at least 4 weeks after the most recent biologic (antibody-based) or immunotherapy ii) at least 2 weeks after any prior chemotherapy or targeted small molecule therapy
* Subjects must have platinum resistant ovarian cancer defined as disease recurrence < 6 months after completion of a platinum-containing regimen. Patients with primary platinum refractory disease are eligible. Primary platinum refractory disease is defined as progression of disease prior to completion of 1st line platinum therapy or immediately following (≤ 3 months following last date of chemotherapy).
* Subjects will have received ≤4 prior lines for platinum resistant ovarian cancer (PROC); maintenance bevacizumab or poly adenosine diphosphate-ribose polymerase (PARP) are not included as a line of therapy.
* Subjects who are eligible for bevacizumab, mirvetuximab, or PARP inhibitor therapy must have received these treatments. For patients who are ineligible for these treatments or those who decline, this must be documented in the records.

Exclusion Criteria:

* Has adverse events (AEs) from prior anti-cancer therapy that have not resolved to Grade ≤ 1, except alopecia.
* Subjects with asymptomatic central nervous system (CNS) metastases are eligible provided they have been clinically stable and not requiring steroid for at least 4 weeks.
* Serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator), such as significant cardiac or pulmonary morbidity e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 3 months.
* Impaired cardiac function or clinically significant cardiac disease.
* Active infection requiring therapy or has a known history of positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody with detected Hepatitis C virus (HCV) RNA. No testing for Hepatitis B or Hepatitis C is required.
* Received a live vaccine within 30 days of planned start of study treatment or requiring a live vaccine during the study.
* Females who are pregnant or breastfeeding.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to paclitaxel.
* Grade 2 peripheral neuropathy at baseline or screening.
* Essential hypertension or any other condition currently being treated with an angiotensin-converting enzyme (ACE)/angiotensin II receptor blockers (ARB) inhibitor, calcium channel blocker, diuretic or any other antihypertensive agent.
* Subjects with a history of orthostasis or syncope.
* Subjects with a history of hypersensitivity, allergy or intolerance to ACE/ARB inhibitors.
* Subjects with baseline systolic blood pressure ≤ 95 or diastolic blood pressure ≤ 60 obtained on two separate days prior to study enrollment.
* Subjects with uncontrolled hypertension at baseline defined as systolic blood pressure ≥ 180 or diastolic blood pressure ≥ 110 on two readings obtained on two separate days prior to study enrollment.
* Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical trial (e.g., substance abuse; psychiatric disturbance; or uncontrolled intercurrent illness including active infection, arterial thrombosis, and symptomatic pulmonary embolism).
* Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results and, in the opinion of the investigator, would make the subject inappropriate for entry into the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Screening through end of treatment, estimated 24 months total.
  ORR will be determined as the number of patients with a partial response (PR) or complete response (CR) to therapy by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Screening through end of treatment, estimated 24 months total
  The time from randomization (or registration) to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation. Response is evaluated using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Oladapo Yeku, MD, Ph.D., FACP, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the Principal Investigator. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation